CLINICAL TRIAL: NCT03497286
Title: Virtual Mentorship to Support Maternal and Infant Health and Wellbeing: Assessing the Impact and Efficacy of NurturePA
Acronym: NPA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Allegheny Singer Research Institute (also known as Allegheny Health Network Research Institute) (Other); University of Michigan (Other)
Responsible Party: Principal Investigator, Lindsay Page, Assistant Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRO17090518
Record Dates: First submitted 2018-04-06; First posted 2018-04-13 (Actual); Last update posted 2021-08-16 (Actual); Status verified 2021-08

CONDITIONS: Mothers
Keywords: maternal health; maternal stress; infant health

STUDY DESIGN:
Intervention Model Description: This study is a randomized control trial design that will compare the outcomes of randomly assigned treatment and control groups after participation in the NurturePA program.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Participants in the treatment condition will be enrolled in the text-based mentorship program and will be able to engage with their assigned mentor as much or as little as they choose.
  Interventions: Behavioral: Text-based mentorship
- Control (Active Comparator): Participants in the control condition will receive periodic informational texts related to the growth and development of their new baby.
  Interventions: Behavioral: Control text messaging

INTERVENTIONS:
Behavioral: Text-based mentorship — The treatment is a text-based peer-to-peer mentorship program for new mothers to promote the healthy development of young children by enhancing the parenting skills of the children's parents. Volunteer mentors who are experienced parents are paired with the parents of newborns. Mentors use text messaging to communicate with, support and encourage new parents while providing best-practice information, answers to the parents' questions, suggestions regarding activities to foster healthy development, and reminders about key milestone activities. The typical NurturePA mentor-mother pair communicates back-and-forth multiple times per week, at any time of the day.
  Arms: Treatment
Behavioral: Control text messaging — Control participants will receive periodic texts from NurturePA with information about child safety and health.
  Arms: Control

SUMMARY:
The primary objective of this study is to determine whether the NurturePA text-based mentorship program reduces maternal stress and depressive symptoms, increases maternal knowledge, and increases engagement in language and literacy practices among new mothers relative to the control condition of periodic informational texts at the four-month data collection point.

DETAILED DESCRIPTION:
Context: New parents in the US are typically offered little if any support with the transition to parenthood, despite the difficulty many families experience during this time and the importance of positive early parent-child interactions to children's future school and life outcomes.

Objectives: This study seeks to evaluate the impact of the NurturePA text-based mentorship program on maternal and infant health and wellbeing.

Study Design: Randomized control trial Setting/Participants: Participants will be recruited from the West Penn Hospital Maternity Ward. 200 participants (100 treatment, 100 control) will be recruited. They must be first or second time mothers of a focal infant of full term gestational age and normal birthweight. They must be current residents of Allegheny County and plan to remain in Allegheny County for the next two years.

Study Interventions and Measures: Treatment participants will be enrolled in the NurturePA text-based mentorship program and assigned a mentor with whom they can communicate. Control participants will receive periodic texts from NurturePA with information about child safety and health.

This study will measure maternal mood and stress, engagement in parent-child language and literacy activities, maternal knowledge, and child developmental outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Resident of Allegheny County
2. First time mother or mother of one other child
3. Gestational age of focal infant at birth is at or above 34 weeks
4. Birthweight of focal infant at or above 4 pounds (1814 grams)
5. Focal infant leaving hospital with mother (e.g. no extended NICU stay)
6. Planning to remain living in Allegheny County for at least two years
7. No more than one other child living full time and being cared for in the home (including non-biological children)

Exclusion Criteria:

1. History of substance abuse disorder
2. Parents/guardians who, in the opinion of the Investigator, may be non-adherent with study schedules or procedures.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 199 (Actual)
Dates: Start 2018-05-09 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Parental Stress | 4 months from study start
  We will measure parental stress using self-administered subscales from the parent domain of the Parenting Stress Index (4th Edition): isolation, attachment, depression, child reinforces parent, and parent competence (15 minutes; Abidin, 2012). As we are omitting subscales that are not of interest, we cannot generate an overall score. Each subscale can be scored individually. Each subscale has a number of items scored 1 (strongly disagree) to 5 (strongly agree). The number of items per subscale and therefore the subscale score ranges vary. The ranges for each subscale are as follows: isolation (6-30), attachment (7-35), depression (9-45), child reinforces parent (6-30), and parent competence (11-55). Subscale scores are calculated by summing each of the responses that correspond with the subscale. Higher scores indicate higher levels of stress, which is considered to be a worse outcome. Percentile scores corresponding to each of the subscale raw scores are also available.
Parental stress | 18 months from study start
  We will measure parental stress at 18 months from study start using two of three self-administered subscales of the Parenting Stress Index Short Form (Fourth Edition): parental distress and parent-child dysfunctional interaction (10 minutes; Abidin, 2012). We will be reporting individual measurements, rather than change over time. As we are omitting subscales that are not of interest to our project, we cannot generate an overall score for the parent domain. However, each subscale can be scored individually. Each subscale has a number of items scored 1 (strongly disagree) to 5 (strongly agree). Each subscale has 12 items and thus score ranges of 12-60. Subscale scores are calculated by summing each of the responses that correspond with the subscale. Higher scores indicate higher levels of stress, which is considered to be a worse outcome. Percentile scores corresponding to each of the subscale raw scores are also available.

SECONDARY OUTCOMES:
Maternal Knowledge | 4 months from study start
  We will adapt the Opinions about Babies questionnaire which was developed by Stephanie Reich as a criterion-referenced knowledge questionnaire for use in a 2005 study (Reich, 2005). The content comes from the Bright Futures Guidelines for Health Supervision, and the American Academy of Pediatrics Guidelines for Health Supervision III (Reich, 2005). It has been used to measure the effects of an educational baby book intervention on maternal knowledge and was shown to be sensitive to intervention effects (Reich et al, 2010). Under the advisement of NurturePA, we selected items that target the types of developmental and self-care knowledge that the program aims to impart. We also edited the wording of some items to more closely target these topics of interest. The edited questionnaire includes 11true/false items. Items are scored 0 if incorrect and 1 if correct and then the items are summed resulting in a final score between 0 and 11. A higher score indicates a better outcome.
Engagement in Language and Literacy Activities | 4 months from study start
  We will measure the mother's level of engagement in activities that support the development of their child's language and literacy activities at 4 months after study start using a self-administered questionnaire. We will report individual scores rather than change over time. The items on the questionnaire are drawn from three sources. Many of the items are taken from a survey administered during the Metro Baby Study, a longitudinal study of low-income minority families in New York City conducted by The Center for Research on Culture, Development, and Education at New York University. Additional items were added based on items from Early Head Start parent surveys and the Ages and Stages 12-month questionnaire (Squires & Bricker, 2009). The 4-month measure will include 8 items scored from 1 (rarely/not at all) to 4 (every day) for a total score range of 8 to 32 where higher scores indicate a better outcome.
Engagement in Language and Literacy Activities | 18 months from study start
  We will measure the mother's level of engagement in activities that support the development of their child's language and literacy activities at 18 months after study start using a self-administered questionnaire. We will report individual scores rather than change over time. The items on the questionnaire are drawn from three sources. Many of the items are taken from a survey administered during the Metro Baby Study, a longitudinal study of low-income minority families in New York City conducted by The Center for Research on Culture, Development, and Education at New York University. Additional items were added based on items from Early Head Start parent surveys and the Ages and Stages 12-month questionnaire (Squires & Bricker, 2009). The 18-month measure will include 11 items scored from 1 (rarely/not at all) to 4 (every day) for a total score range of 11 to 44 where higher scores indicate a better outcome.
Child Development | 4 months from study start
  We will measure child development at 4 months after study start using a self-administered questionnaire asking mothers to report whether their baby has reached particular developmental milestones. We will report individual scores rather than change over time. At 4 months after study start the questionnaire will include 5 items scored from 1 (not yet) to 3 (yes) for a total score range of 5 to 15 where higher scores indicate a better outcome.
Child Development | 18 months from study start
  We will measure child development at 18 months after study start using a self-administered questionnaire asking mothers to report whether their baby has reached particular developmental milestones. We will report individual scores rather than change over time. At 18 months after study start the questionnaire will include 10 items scored from 1 (not yet) to 3 (yes) for a total score range of 10 to 30 where higher scores indicate a better outcome.
WIC Usage | 4 and 18 months from study start
  We will measure WIC usage at 4 months after study start and 18 months after study start by using data from the Allegheny County Integrated Data Systems. WIC usage will be measured in the length of time receiving WIC benefits.
Early Language and Development Screening | 4 and 18 months from study start
  We will measure usage of early language and development screening services 4 months after study start and 18 months after study start by using data from the Allegheny County Integrated Data Systems. Screening usage will be measured with a binary indicator of whether or not a mother has used screening services.
Edinburgh Postnatal Depression Scale | 4 months from start of the study
  This is a 10-question self-rating scale for assessing perinatal depression. The scale is administered at approximately 4 months post-partum during the course of a well-baby doctor's office visit. Each of the 10 items is scaled on a 0-3 scale and then these item scores are summed for an overall score. Overall scores are interpreted as follows: 0-8 (low probability of depression); 8-12 (most likely just dealing with a new baby or the baby blues); 13-14 (signs leading to possibility of post-partum depression); 15+ (high probability of experiencing clinical depression).

CONTACTS AND LOCATIONS:
Overall Officials: Lindsay C Page, Ed.D., Principal Investigator — University of Pittsburgh; Christina Weiland, Ed.D., Principal Investigator — University of Michigan
Locations (1):
- West Penn Hospital, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
A full de-identified participant level data file will be available for future studies.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available for request upon publication of results from this study.
Access Criteria: Interested researchers will need to seek permission through the clinical site IRB and the study PI. Interested researchers will need to enter into a data use agreement with the Allegheny-Singer Research Institute.

REFERENCES:
- See also: NurturePA is the non-profit organization which runs the text-based mentorship program for new mothers that we are investigating. — http://nurturepa.org/